CLINICAL TRIAL: NCT05336942
Title: Effects of Mild Cognitive Impairment on Auditory System and Its Correlation With Cognitive Function: a Multicenter, Randomized Controlled Study
Brief Title: Correlation Between Prognosis of Mild Cognitive Impairment and Hearing Function in Community Elderly
Status: Completed | Type: Observational
Sponsor: Tongji University (Other)
Responsible Party: Principal Investigator, Jie Tong, Professor, Tongji University
Other Study IDs: PKJ2019-Y24
Record Dates: First submitted 2022-04-09; First posted 2022-04-20 (Actual); Last update posted 2022-04-20 (Actual); Status verified 2022-04

CONDITIONS: Mild Cognitive Impairment
Keywords: mild cognitive impairment; auditory; cognitive function
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- MCI-HI group: Mild cognitive impairment and hearing impairment group
- MCI-nHI group: Mild cognitive impairment and no hearing impairment group
- Control group: Control group

SUMMARY:
Cognitive dysfunction is a high incidence disease in the elderly. To date, there is no effective treatment. At the same time, early cognitive impairment is easy to be ignored, delayed intervention. Most patients develop moderate or severe dementia with hearing loss before treatment. At present, there are few studies on the correlation between mild cognitive impairment and hearing function. The investigators evaluated CDR, MMSE, MoCa, and hearing tests at baseline, 6 months later, and 12 months later in a multicenter, randomized cohort study of adults aged 55-65 years. To investigate the correlation between mild cognitive impairment and hearing impairment and its possible predictors. The investigators hope to provide more evidence-based evidence for early identification of mild cognitive impairment.

DETAILED DESCRIPTION:
With the aging of society, the health of the elderly has paid more and more attention. Cognitive dysfunction has always been a common disease that seriously affects the quality of life of the elderly, thus increasing the burden of family and society. How to prevent and slow down cognitive dysfunction is a topic worthy of discussion, but so far, there is no safer and effective method to solve this problem.

Cognitive function refers to various conscious mental activities of human beings in the state of awakening, including reception function, namely receiving external information through various senses, memory and learning function, thinking function and expression function. Mild cognitive impairment (MCI) is the early stage of Senile dementia and a cognitive loss state between normal aging and dementia. The reception function of sensory organs is the basis of the whole cognitive activity and the initial stage of cognitive function, so there is a close relationship between sensation and cognitive function. Studies have shown that hearing impairment is an independent risk factor for cognitive impairment, hearing loss is positively correlated with cognitive impairment, and senile MCI is significantly correlated with hearing impairment, both of which exist a dose-effect relationship and complement each other. Especially in people over 50 years old, hearing impairment has a high incidence of cognitive impairment, and hearing impairment is an influential factor of cognitive function. There is a certain correlation between hearing loss and cognitive function. Bai Jie et al. analyzed the MMSE, MoCA, drawing clock test and daily living ability Assessment Scale of the normal hearing group and the untreated senile deafness group, and showed that hearing loss would lead to cognitive impairment, mainly for two reasons: (1) People with presbyopia do not have a good understanding of the tasks to be performed; (2) Presbyopia causes social isolation and cognitive decline.

American Medical Association (ASA) study included 1,884 subjects, of whom 1,162 had presbyage-related deafness, and the results showed that these patients had lower cognitive function than normal hearing subjects. They believe that the reason is that both senile deafness and cognitive decline occur in the same neural source. Therefore, it is worth exploring whether cognitive function can be delayed and improved by improving hearing. There are a large number of people over 60 years old with hearing impairment. According to the Chinese Epidemiological survey, 35-55% of people over 60 years old suffer from different degrees of hearing impairment. But as most of the older hearing impairment is a process of gradual development, thus can be considered as a immutable physiological process, and this is a kind of don't want to expose himself, and is hard to see someone invisible disability, therefore, are easily ignored by others, resulting in social communication, interpersonal communication between the obstacle, thus reducing the social function of old people.

To date, there are few prospective studies on the relationship between hearing impairment and cognitive impairment. This research through the community elderly were followed up for 1 year, evaluation of hearing loss and the correlation between prognosis of mild cognitive function impairment, focus on community elderly hearing impairment and the relationship between the cognitive dysfunction, to strengthen the science popularization of the old man, so that more older people can focus on listening and impaired cognitive function, active intervention, In this way, the quality of life of the elderly can be improved, social communication can be promoted, life satisfaction of the elderly can be improved, and family and social burden can be reduced.

ELIGIBILITY:
Inclusion Criteria:

1. The registered residence of local residents is more than one month.
2. Aged 55 to 65 years.
3. Be able to conduct verbal communication or written conversation, or complete the investigation with the help of family members.

Exclusion Criteria:

1. Mini-mental state examination(MMSE), illiterate group ≤ 17 points, primary school group ≤ 20 points, middle school or above group 24 points;
2. Those who meet the ICD-10 diagnostic criteria for dementia;
3. Those who are obviously blind or have difficulty in speech expression;
4. Persons suffering from serious physical diseases;
5. Those who meet the diagnostic criteria of schizophrenia, neurosis, organic mental disorder and mental retardation;
6. Persons with severe or above hearing impairment;
7. Those who are unable to sign the informed consent form.

Ages: 55 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mild cognitive impairment in the community
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-12-30 (Actual); Study Completion 2022-03-30 (Actual)

PRIMARY OUTCOMES:
Mini-mental state examination (MMSE) | Baseline
  To screen and assess the extent of cognitive dysfunction.
Mini-mental state examination (MMSE) | 6-month
  To screen and assess the extent of cognitive dysfunction.
Mini-mental state examination (MMSE) | 12-month
  To screen and assess the extent of cognitive dysfunction.
Montreal Cognitive Assessment (MocA) | Baseline
  To evaluate various domains of cognition.
Montreal Cognitive Assessment (MocA) | 6-month
  To evaluate various domains of cognition.
Montreal Cognitive Assessment (MocA) | 12-month
  To evaluate various domains of cognition.
Pure tone Listening Test (PTA) | Baseline
  To determine the threshold intensity of hearing at each frequency and measure the nature and extent of hearing loss.
Pure tone Listening Test (PTA) | 6-month
  To determine the threshold intensity of hearing at each frequency and measure the nature and extent of hearing loss.
Pure tone Listening Test (PTA) | 12-month
  To determine the threshold intensity of hearing at each frequency and measure the nature and extent of hearing loss.

SECONDARY OUTCOMES:
Clinical Dementia Rating (CDR) | Baseline
  To generated to stage the severity of dementia.
Clinical Dementia Rating (CDR) | 6-month
  To generated to stage the severity of dementia.
Clinical Dementia Rating (CDR) | 12-month
  To generated to stage the severity of dementia.
Auditory brainstem response (ABR) | Baseline
  To evaluate objectively the hearing level by the response threshold of V wave.
Auditory brainstem response (ABR) | 6-month
  To evaluate objectively the hearing level by the response threshold of V wave.
Auditory brainstem response (ABR) | 12-month
  To evaluate objectively the hearing level by the response threshold of V wave.

CONTACTS AND LOCATIONS:
Overall Officials: Jie Yuan, M.D., Principal Investigator — Tongji University
Locations (1):
- Tongji University, Shanghai, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Srikanth V, Sinclair AJ, Hill-Briggs F, Moran C, Biessels GJ. Type 2 diabetes and cognitive dysfunction-towards effective management of both comorbidities. Lancet Diabetes Endocrinol. 2020 Jun;8(6):535-545. doi: 10.1016/S2213-8587(20)30118-2. PMID 32445740
- [Result] Ringman JM, Medina LD, Rodriguez-Agudelo Y, Chavez M, Lu P, Cummings JL. Current concepts of mild cognitive impairment and their applicability to persons at-risk for familial Alzheimer's disease. Curr Alzheimer Res. 2009 Aug;6(4):341-6. doi: 10.2174/156720509788929336. PMID 19689233
- [Result] Heywood R, Gao Q, Nyunt MSZ, Feng L, Chong MS, Lim WS, Yap P, Lee TS, Yap KB, Wee SL, Ng TP. Hearing Loss and Risk of Mild Cognitive Impairment and Dementia: Findings from the Singapore Longitudinal Ageing Study. Dement Geriatr Cogn Disord. 2017;43(5-6):259-268. doi: 10.1159/000464281. Epub 2017 Apr 19. PMID 28420004
- [Result] Jongsiriyanyong S, Limpawattana P. Mild Cognitive Impairment in Clinical Practice: A Review Article. Am J Alzheimers Dis Other Demen. 2018 Dec;33(8):500-507. doi: 10.1177/1533317518791401. Epub 2018 Aug 1. PMID 30068225
- [Result] Maharani A, Pendleton N, Leroi I. Hearing Impairment, Loneliness, Social Isolation, and Cognitive Function: Longitudinal Analysis Using English Longitudinal Study on Ageing. Am J Geriatr Psychiatry. 2019 Dec;27(12):1348-1356. doi: 10.1016/j.jagp.2019.07.010. Epub 2019 Jul 22. PMID 31402088
- [Result] Lin FR, Yaffe K, Xia J, Xue QL, Harris TB, Purchase-Helzner E, Satterfield S, Ayonayon HN, Ferrucci L, Simonsick EM; Health ABC Study Group. Hearing loss and cognitive decline in older adults. JAMA Intern Med. 2013 Feb 25;173(4):293-9. doi: 10.1001/jamainternmed.2013.1868. PMID 23337978
- [Result] Khan HZ, Park CY, Lim MA, Beltran AJ, Farquhar D, Yencha M, Capra GG. Radiographic findings in young adults with asymmetric sensorineural hearing loss. Am J Otolaryngol. 2019 Jan-Feb;40(1):78-82. doi: 10.1016/j.amjoto.2018.10.003. Epub 2018 Oct 11. PMID 30472122
- [Derived] Tong J, Zhang J, Xu L, Liu M, Min J, Yao M, Cheng X, Zhang Q, Sun X, Yuan J. Effect of hearing loss on cognitive function in patients with mild cognitive impairment: A prospective, randomized, and controlled study. Front Aging Neurosci. 2022 Aug 1;14:934921. doi: 10.3389/fnagi.2022.934921. eCollection 2022. PMID 35978946